CLINICAL TRIAL: NCT04795141
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Tolerability of ABY-035 in the Treatment of Subjects With Ankylosing Spondylitis
Brief Title: ABY-035 in the Treatment of Subjects With Ankylosing Spondylitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor's development strategy is adjusted.
Sponsor: Inmagene LLC (Industry)
Collaborators: Affibody (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABY-035-204
Record Dates: First submitted 2021-03-03; First posted 2021-03-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- #1: Cohort 1-High Dose Q2W (Experimental): Cohort 1: ABY-035 High Dose, every 2 weeks, subcutaneous injection
  Interventions: Drug: ABY-035
- #2: Cohort 1-High Dose Q4W (Experimental): Cohort 1: ABY-035 High Dose, every 4 weeks, subcutaneous injection
  Interventions: Drug: ABY-035
- #3: Cohort 1-Low Dose Q2W (Experimental): Cohort 1: ABY-035 Low Dose, every 2 weeks, subcutaneous injection
  Interventions: Drug: ABY-035
- #4: Cohort 2-Low Dose QW (Experimental): Cohort 2: ABY-035 Low Dose, every week, subcutaneous injection
  Interventions: Drug: ABY-035
- #5: Cohort 2-High Dose QW (Experimental): Cohort 2: ABY-035 High Dose, every week, subcutaneous injection
  Interventions: Drug: ABY-035
- #1: Cohort 1-Placebo Q2W (Placebo Comparator): Cohort 1: Placebo, every 2 weeks, subcutaneous injection
  Interventions: Drug: Placebo
- #2: Cohort 2-Placebo QW (Placebo Comparator): Cohort 2: Placebo, every week, subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABY-035 — ABY-035 Solution for injection
  Other Names: Izokibep
  Arms: #1: Cohort 1-High Dose Q2W; #2: Cohort 1-High Dose Q4W; #3: Cohort 1-Low Dose Q2W; #4: Cohort 2-Low Dose QW; #5: Cohort 2-High Dose QW
Drug: Placebo — Normal Saline for injection
  Other Names: Normal Saline
  Arms: #1: Cohort 1-Placebo Q2W; #2: Cohort 2-Placebo QW

SUMMARY:
ABY-035-204 is a clinical study to assess the efficacy of IL-17 blocker ABY-035 in ankylosing spondylitis(AS). The primary objective is to estimate the relationship between different dose regimens of ABY-035 and clinical response as assessed by Assessment of Spondyloarthritis International Society 40 (ASAS40) response at Week 16 in subjects with active AS.

DETAILED DESCRIPTION:
ABY-035-204 is a double-blind, randomized, parallel-group, placebo-controlled study.

The primary objective is to estimate the relationship between different dose regimens of ABY-035 and clinical response as assessed by Assessment of Spondyloarthritis International Society 40 (ASAS40) response at Week 16 in subjects with active AS.

The study will include the following 3 periods:

1. Screening Period: Up to 35 days prior to baseline randomization.
2. Treatment Period 1: Day 0-Week 16

   Cohort 1: Eligible subjects will be randomized 1:1:1:1 to receive 1 of 4 treatments (ABY-035 High Dose every 2 weeks (Q2W), ABY-035 Low Dose every 2 weeks (Q2W), ABY-035 High Dose every 4 weeks (Q4W), or placebo Q2W), and will remain on their allowable background medication.

   Cohort 2: Eligible subjects will be randomized 1:1:1 to receive 1 of 3 treatments (ABY-035 High Dose every week (QW), ABY-035 Low Dose every week (QW), or placebo QW), and will remain on their allowable background medication.

   Randomization will be stratified by region (North Eastern Asia and North America) and previous tumor necrosis factor alpha (TNFα) inhibitor exposure (TNFα inhibitor treated or TNFα inhibitor naïve). Maximum 30% of subjects will be TNFα inhibitor-treated subjects to ensure a representative population for the assessment of efficacy and safety.

   Treatment Period 1 ends at Week 16 after all trial assessments have been done and Treatment Period 2 starts at Week 16 with the IMP injection.
3. Treatment Period 2 (Extension Period): Week 16-Week 52 Cohort 1: Subjects will receive ABY-035 High Dose Q2W treatment in an open-label manner.

Cohort 2: Subjects will receive ABY-035 High Dose QW treatment in an open-label manner.

At Week24, subjects who could not achieve an ASAS20 response from baseline are defined as non-responders and will discontinue the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years of age.
2. Subjects with active AS, determined by documented radiologic evidence (X-ray) fulfilling the Modified New York criteria for AS (1984).

   AND At least one SpA feature, according to ASAS criteria.
3. Subjects have moderate to severe active disease
4. Subjects must have inadequate response or intolerance to at least 2 NSAIDs, or contraindication to NSAID therapy.
5. Subjects may be TNFα inhibitor-naïve or may have received up to 2 prior TNFα inhibitor(s)..

Exclusion Criteria:

1. Subjects have active fibromyalgia or total spinal ankylosis ('bamboo spine'), or any other inflammatory arthritis.
2. Subjects have used medications in the manner as detailed by the exclusion criteria as detailed in the study protocol.
3. Subjects have received technetium-99 conjugated with methylene diphosphonate other than for diagnostic purpose within 5 years prior to baseline.
4. Have received any live (includes attenuated) vaccination within the 12 weeks prior to the baseline.
5. Subjects have received any non-biological therapy for AS not listed as detailed in the study protocol within or outside a clinical study in the 3 months or within 5 half-lives prior to the Baseline Visit (whichever is longer).
6. Subject has an active infection or history of infections
7. Have evidence of or test positive for hepatitis B virus (HBV)
8. Have evidence of or test positive for hepatitis C virus (HCV).
9. Have a historically positive human immunodeficiency virus (HIV) test or test positive at screening for HIV.
10. Subjects have known tuberculosis (TB) infection, at high risk of acquiring TB infection, or current or history of nontuberculous mycobacterium (NTMB) infection, or LTB.
11. Have a history of a lymphoproliferative disorder including lymphoma or current signs and symptoms suggestive of lymphoproliferative disease.
12. Subjects have active Crohn's disease (CD) or active ulcerative colitis (UC).
13. Subjects have active uveitis within 6 weeks prior to baseline.
14. Subjects have laboratory abnormalities at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving an ASAS40 response | 16 weeks
  The treatment effect

SECONDARY OUTCOMES:
Change from baseline in BASDAI | 16 weeks
  The treatment effect
Change from baseline in BASFI | 16 weeks
  The treatment effect
Proportion of subjects reaching ASDAS-MI | 16 weeks
  The treatment effect
Incidence of AEs | 74 weeks
  Safety information
Incidence of serious adverse events (SAEs) and adverse events of special interests (AESIs) | 74 weeks
  Safety information
AEs leading to withdrawal from investigational medicinal product (IMP) | 74 weeks
  Safety information
Change in safety laboratory parameters and vital signs compared to baseline | 74 weeks
  Safety information
Proportion of subjects achieving an ASAS40 response, ASAS20 response, ASAS partial remission, and ASAS 5/6 response respectively at required timepoints | 52 weeks
  The treatment effect
Change from baseline in BASDAI and BASFI at required timepoints | 52 weeks
  The treatment effect
Proportion of subjects reaching BASDAI50 and ASDAS-MI at required timepoints | 52 weeks
  The treatment effect
Proportion of subjects experiencing clinically important improvement at required timepoints | 52 weeks
  The treatment effect
ASDAS-CRP and ASDAS status at required timepoints | 52 weeks
  The treatment effect
Change from baseline in total and nocturnal pain at required timepoints | 52 weeks
  The treatment effect

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence He, Study Director — SVP, Global Regulatory Head
Locations (47):
- United States (15):
  - Arizona Arthritis & Rheumatology Research, PLLC, Glendale, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Newport Huntington Medical Group, Huntington Beach, California
  - Desert Medical Advances, Palm Desert, California
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Drucker Sarasota Arthritis Research Center, Sarasota, Florida
  - Greater Chicago Specialty Physicians/ Clinical Investigation Specialists, Inc., Schaumburg, Illinois
  - Clinic of Robert Hozman, MD / Clinical Investigation Specialists,, Skokie, Illinois
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - M3 Emerging Medical Research, LLC, Durham, North Carolina
  - Clinical Research Source, Inc., Perrysburg, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - HRMD Research, Dallas, Texas
  - Seattle Rheumatology Associates, Seattle, Washington
- China (25):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Chao-Yang Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Sun Yat-Sen Memorial Hospital Sun Yat-Sen University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tong Ji Hospital TongJi Medical Colleague of HUST, Wuhan, Hubei
  - Zhuzhou Hospital Affiliated to Xiangya School of Medicine, Zhuzhou, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and TechNology, Baotou, Inner Mongolia
  - The Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Linyi People's Hospital, Linyi, Shandong
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Kaohsiung Chang Gung Memorial Hospital ，Chang Gung Medical Foundation, Gaoxiong, Taiwan
  - Kaohsiung Veterans General Hospital, Gaoxiong, Taiwan
  - National Taiwan University Hospital (NTUH), Taibei, Taiwan
  - Tri-Service General Hospital, Taibei, Taiwan
  - China Medical University Hospital (CMUH), Taizhong, Taiwan
  - Chung Shan Medical University Hospital (CSMHU), Taizhong, Taiwan
  - The Affiliated Hospital of The Affiliated Hospital of Inner Mongolia Medical University Medical University, Hohhot, The Affiliated Hospital of Inner Mongolia Medical University
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
- South Korea (7):
  - Chonnam National University Hospital, Gwangju, Gwangju
  - Ajou University Hospital, Gyeonggi-do
  - Bundang Seoul National University Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Hanyang University Seoul Hospital, Seoul
  - Kyunghee University Hospital, Seoul
  - SNU Boramae Medical Center, Seoul